CLINICAL TRIAL: NCT00920634
Title: Protocol for Drug Use Investigation of Follistim Injection
Brief Title: Protocol for Drug Use Investigation of Follistim Injection (Study P06132)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P06132
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Anovulation
MeSH Terms: conditions — Anovulation | interventions — follitropin beta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with anovulation and oligoovulation due to hypothalamus-pituitary dysfunction (amenorrhea first grade, anovulatory cycle, polycystic ovary syndrome, oligoamenorrhea) who underwent ovulation induction
  Interventions: Drug: Follitropin beta

INTERVENTIONS:
Drug: Follitropin beta — For subcutaneous or intramuscular injection, the usual dosage is 50 IU of follitropin beta (recombinant) once daily for 7 days. The dosage should be adjusted subsequently while monitoring the development of follicles (dose increase by 25 IU every 7 days if the response of the ovaries is poor) and, after confirming presence of follicles of 18 mm or larger in mean diameter by the ultrasonic tomography, ovulation is induced by the administration of a human chorionic gonadotropin preparation.

SUMMARY:
The main purpose of this investigation is to collect information about safety and efficacy of Follistim Injection from actual clinical use to induce ovulation in patients with anovulation and oligoovulation due to hypothalamus-pituitary dysfunction.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent IVF

Exclusion Criteria:

* Patients with tumors of ovary, breast, uterus, pituitary or hypothalamus
* Pregnant or possible pregnant women, or lactating women
* Patients with undiagnosed atypical vaginal bleeding
* Patients with a history of hypersensitivity to any of the ingredients of this product
* Patients with ovarian cysts or enlarged ovaries, not related to polycystic ovarian disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese 300 patients
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of ovulation | 3 months, from initiation of treatment to confirmation of pregnancy.

SECONDARY OUTCOMES:
Pregnancy outcome | 3 months, from initiation of treatment to confirmation of pregnancy.